CLINICAL TRIAL: NCT01195402
Title: Low Intensity Pulmonary Outpatient Rehabilitation in Moderate to Severe COPD
Brief Title: Ambulatory Interdisciplinary Rehabilitation in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: AIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Dr. Tibor Schmoller, pulmonary practice Winterhude (Unknown)
Responsible Party: Dr. Andreas Meyer, Kliniken Mariahilf GmbH, Department of Pneumology, Mönchengladbach, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIR-01
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: COPD
Keywords: COPD; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Subjects do not receive any kind of active intervention.
- pulmonary outpatient rehabilitation (Active Comparator): Subjects participate in an outpatient pulmonary rehabilitation program
  Interventions: Procedure: pulmonary outpatient rehabilitation

INTERVENTIONS:
Procedure: pulmonary outpatient rehabilitation — Subjects take part in once weekly training sessions of 60 min duration. Sessions take place in local physiotherapist practice and involve simple training devices (chairs, elastic bands, balls). In addition, subjects take part in a structured and validated educational program concerning COPD (COBRA) of 8 h duration. They are offered counselling regarding nutrition (2 h), psycho-social (2 h) and social (2 h) aspects.
  Arms: pulmonary outpatient rehabilitation

SUMMARY:
This randomised-controlled study is undertaken to investigate the effects of a long term low intensity outpatient training program on physical fitness and quality of life in moderate to severe COPD patients.

DETAILED DESCRIPTION:
Broad evidence exists on the beneficial effects of pulmonary rehabilitation on exercise capabilities and quality of life in COPD patients. Clinically relevant effects have been achieved by training programs of differing design regarding setting (inpatient vs. outpatient vs. home-based), duration (short-term vs. long-term) and intensity (high vs. low intensity).

While there is sufficient evidence to propose pulmonary rehabilitation its use is generally low in clinical practice. One reason may be that it is unlikely that costly programs are offered to a significant proportion of eligible patients. The ideal training program will therefore at the same time accomplish the greatest improvements regarding physical capabilities and quality of life and sustain them for the longest period at the lowest cost.

The purpose of the present study is to evaluate whether a continuous, low-intensity, low-cost, physiotherapist-led outpatient pulmonary rehabilitation program is a able to achieve significant long-term improvements of exercise tolerance and quality of life in moderate to severe COPD patients at a lower cost level than previously published programs.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD stage II-IV
* smoking history of >20 pack years
* adequate pharmacological therapy
* written informed consent

Exclusion Criteria:

* respiratory insufficiency, defined as PaO2<55 mm Hg and/or PaCO2>50 mm Hg breathing room air
* manifest cardiac insufficiency
* uncontrolled arterial hypertension
* malignant disease
* symptomatic coronary heart disease resp. pathological cycle ergometry results
* limited physical capabilities caused by musculoskeletal disorders
* unwillingness to return for follow-up
* previous or ongoing participation in exercise training programs
* unability to attend at least 75% of sessions

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-04; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
6-Minute walk distance | Six months

SECONDARY OUTCOMES:
Quality of life | Six months
  General and disease-specific health-related quality of life measured using the Short-Form 36-Questionaire resp. the St. George's-Respiratory Questionaire
Maximum oxygen uptake | Six months
  Maximum oxygen uptake measured during unsteady state cycle ergometer test with work increments of 10 watts each minute until exhaustion.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meyer, M.D., Principal Investigator — Kliniken Mariahilf GmbH, Mönchengladbach, Germany
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Baumann HJ, Kluge S, Rummel K, Klose H, Hennigs JK, Schmoller T, Meyer A. Low intensity, long-term outpatient rehabilitation in COPD: a randomised controlled trial. Respir Res. 2012 Sep 27;13(1):86. doi: 10.1186/1465-9921-13-86. PMID 23017153